CLINICAL TRIAL: NCT00237900
Title: An Open, Single.Centre, Phase I/II Study of ZD1839 (Iressa) in Combination With 5-Fluorouracil, Leucovorin and Radiotherapy in Subjects With Resectable Gastric Cancer
Brief Title: Gefitinib in Combination With Chemoradiation in Resectable Gastric Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0539
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Subjects With Resectable Local or Locally Advanced, Non-Metastatic (T2-T4, N0-N3, M0; Stages II and III) and Histologically-Confirmed Intestinal GC
MeSH Terms: interventions — Gefitinib; Fluorouracil; Leucovorin; Radiotherapy

INTERVENTIONS:
Drug: Gefitinib, 5-fluorouracil, leucovorin and radiotherapy

SUMMARY:
To assess safety, efficacy and explorative objectives of gefitinib in combination with chemoradiation in resectable gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed intestinal GC (T2-T4)
* Local or locally advanced stage II or stage III gastric cancer of an upper part of the stomach or GE junction
* Lymph node positive or negative
* Metastasis negative
* Resection with curative intent (R0, D2)
* Chemo- and radiotherapy naïve
* Measurable lesion according RECIST
* Written informed consent

Exclusion Criteria:

* Aged below 45 or over 70
* Prior gastric surgery
* Active ILD

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2003-07; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety and tolerability of gefitinib 250 mg in combination with radiotherapy (incidence of DLTs)
Parts 2 and 3: Safety and tolerability of gefitinib in combination with 5-FU, LV and radiotherapy

SECONDARY OUTCOMES:
Parts 2 and 3:
Objective tumour response rate a week before surgery (CR and PR, RECIST criteria).
Objective histological response rate in dissected GC specimens taken at surgery, estimated using Evans/Pisters scores
Exploratory outcome: Parts 2 and 3: sVEGF levels, EGFR activation, Biomarkers such as cyclin D1, IL-1, GI-associated TOP2A, GAS, EST AA552509

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (1):
- Reseach Site, Helsinki, Finland